CLINICAL TRIAL: NCT00534625
Title: Phase 2 Study of the Assessment of Pulmonary Function, Safety, Tolerability, and PK of Zileuton Injection in Patients With Chronic Stable Asthma
Brief Title: Assessment of PFT, Safety, and PK of Zileuton Injection in Asthma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Critical Therapeutics (Industry)
Responsible Party: Cornelis Wortel MD, PhD/Acting CMO, Clinquest Inc
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTI-04-C07-202
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2008-03-21 (Estimated); Status verified 2008-03

CONDITIONS: Asthma
Keywords: Asthma, exacerbation, pulmonary function
MeSH Terms: conditions — Asthma | interventions — zileuton

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator)
  Interventions: Drug: placebo
- 2 (Experimental): 150 mg zileuton by intravenous injection
  Interventions: Drug: zileuton
- 3 (Experimental): 300 mg zileuton by intravenous injection
  Interventions: Drug: zileuton

INTERVENTIONS:
Drug: zileuton — Single injection of zileuton 150 mg
  Arms: 2
Drug: placebo — Single injection of placebo
  Arms: 1
Drug: zileuton — Single injection of zileuton 300 mg
  Arms: 3

SUMMARY:
A single intravenous injection of zileuton (150 or 300 mg) will be administered to patients with stable asthma. The goals will be to determine if zileuton i.v. can produce a rapid increase in FEV1/PEFR and when this effect can be seen. The safety of this route of administration of zileuton will also be studied. PK will be obtained in a population based method.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 12 years of age or older
2. Diagnosis of asthma by current ATS guidelines
3. FEV1 of 4-80%.
4. Reversibility of at least 13% after bronchodilator treatment
5. Must be willing to with hold SABA for 6 hours and ICS for 24 hours prior to treatment.
6. Informed consent

Exclusion Criteria:

1. Females of child bearing potential unless using birth control
2. Uncontrolled systemic disease
3. Known hypersensitivity to zileuton or components of zileuton injection.
4. Upper or lower respiratory tract infection within the last 2 weeks
5. Admission to hospital or ER visit for asthma exacerbation within the last 3 months
6. Course of oral or parenteral steroids within the last 3 months
7. Current smoker or H/O > 15 pack years
8. Creatinine > 1.5 x ULN
9. ALT > 3 x ULN
10. BP < 100 (systolic)
11. H/O HIV
12. H/O alcohol or drug abuse
13. Patients taking Xolair, theophylline, montelukast, zafirlukast, nedocromil, cromolyn sodium, Zyflo (within the past 7 days), warfarin, propranolol, inhaled anti-cholinergics, or LABA.
14. Pregnant or breast feeding females
15. Current participation or participation in an experimental drug study within 30 days.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-09; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Effect on pulmonary function | Within 0-12 hours after single dose

SECONDARY OUTCOMES:
Safety assessments | Within 0-36 hours after single dose

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Cees Wortel, Study Director — Critical Therapeutics